CLINICAL TRIAL: NCT01468324
Title: Phase I Trial of AZD7451, A Topomysin-Receptor Kinase (TRK) Inhibitor, For Adults With Recurrent Glioblastoma Multiforme (GBM)
Brief Title: AZD7451 for Recurrent Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120005; 12-C-0005
Record Dates: First submitted 2011-11-05; First posted 2011-11-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-04-22

CONDITIONS: Glioblastoma Multiforme
Keywords: Brain; Angiogenesis; Radiotherapy; Malignant; Tumor; Glioma; Glioblastoma Multiforme; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Neoplasms; Glioma; Brain Neoplasms | interventions — AZD7451

INTERVENTIONS:
Drug: AZD7451 — Depending on dose level, AZD7451 will be given once daily for 28 day cycles.

SUMMARY:
Background:

- AZD7451 is a drug that may help interfere with brain tumor cell growth. It can prevent glioma cells from entering into normal brain tissue, and slow or stop the growth of additional tumors. Researchers want to see if AZD7451 is effective against gliomas that have not responded to surgery, radiation, or chemotherapy.

Objectives:

- To see if AZD7451 is a safe and effective treatment for gliomas that have not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have gliomas that have not responded to standard treatments.

Design:

* Participants will be screened with a physical exam, medical history, blood and urine tests, heart function tests, an eye exam, and imaging studies.
* Participants will take AZD7451 daily by mouth for 28-day cycles of treatment.
* Participants will keep a medication diary and record any side effects. Treatment will be monitored with frequent blood tests and imaging studies.
* Treatment will continue as long as there are no serious side effects and the tumor does not start growing again....

DETAILED DESCRIPTION:
BACKGROUND:

Recurrent glioma patients have very limited treatment options. A major cause of gliomarelated morbidity and mortality is the extensive infiltrative and invasive nature of glioma cells. Thus, inhibition of glioma invasion is a potentially promising strategy.

Work in the Neuro-Oncology Branch laboratory of Dr. Howard Fine has identified TrkA as an important signaling receptor for mediating glioma cell invasion. Both genetic and pharmacological inhibition of Trk potently inhibits glioma invasion and tumor progression in vitro and in vivo. AZD7451 is a first in-class inhibitor of Trk.

OBJECTIVES:

To establish the maximally tolerated dose (MTD) of continuous twice a day AZD7451 dosing in patients with recurrent glioblastoma not on enzyme-inducing anti-epileptic drugs (EIAED).

To generate pharmacokinetic data on continuous twice a day AZD7451 dosing.

ELIGIBILITY:

Patients with histologically proven glioblastoma are eligible for this study. Patients should have failed prior standard treatment with radiotherapy.

DESIGN:

This study will accrue up to 60 evaluable patients. Cohorts of 3 to 6 patients will receive continuous AZD7451 twice a day orally for 28 days. The MTD will be based on the tolerability observed during the first 4 weeks of treatment only. Up to three patients may be enrolled simultaneously at each dose level. The dose of AZD7451 can be progressively escalated if only 0/3 or 1/6 patients experience a dose limiting toxicity at the prior dose level.

At the end of Cycle 1, patients may choose to continue to receive AZD7451 until disease progression or until they experience unmanageable drug related toxicity, as long as they are continuing to derive clinical benefit and do not fulfill any of the criteria for removal from protocol therapy. Each cycle during this extension period will last 28 days.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically proven malignant primary gliomas who have progressive disease after radiotherapy will be eligible for this protocol.
* Patients must have an MRI scan performed within 14 days prior to registration and on a fixed dose of steroids for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MRI is required.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  1. Patients will be eligible four weeks after surgery if they have recovered from the effects of surgery.
  2. Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease postoperatively, an MRI should be done:
* no later than 96 hours in the immediate post-operative period or
* at least 4 weeks post-operatively, and
* within 14 days of registration, and
* on a stable steroid dosage for at least 5 days.

If the 96 hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required on a stable steroid dosage for at least 5 days.

* Patients must have failed prior radiation therapy.
* Ability of subject or Legally Authorized Representative (LAR) (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of this study.
* Patients must be greater than or equal to18 years old, and must have a life expectancy > 8 weeks. Because no dosing or adverse event data are currently available on the use of AZD7451 in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Patients must have a Karnofsky performance status of greater than or equal to 60
* Patients must be at least 4 weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide, 3 weeks from procarbazine, 2 weeks from vincristine and 2 weeks from last bevacizumab administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents. With the exception of alopecia, all toxicities from prior therapies should be resolved to CTCAE less than or equal to grade 1.
* Patients must have adequate bone marrow function (WBC greater than or equal to 3,000/microl, ANC greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to 9 gm/dl), adequate liver function (AST, ALT and alkaline phosphatase less than or equal to 2.5 times ULN and bilirubin less than or equal to 1.5 times ULN), and adequate renal function (creatinine less than or equal to 1.5 times ULN and/or creatinine clearance greater than or equal to 50 cc/min calculated by Cockcroft-Gault) before starting therapy. Patients must also have serum potassium greater than or equal to 3.5 mmol/L, magnesium, phosphate and calcium levels within normal levels; supplementation is allowed. In cases where the serum calcium is below the normal range, 2 options would be available: 1) the calcium adjusted for albumin is to be obtained and substituted for the measured serum value. Exclusion is to then be based on the adjusted for albumin values falling below the normal limit. 2) Determine the ionized calcium levels. Exclusion is then to be based on whether these ionized calcium levels are out of normal range despite supplementation. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
* Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.
* The effects of AZD7451 on the developing human fetus are unknown. For this reason and because AZD7451 is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or herpartner is participating in this study, the treating physician should be informed immediately.
* A 12 lead electrocardiogram (ECG) to be performed within 2 weeks of trial entry with QTc less than or equal to 470 msec.
* Patients must have normal left ventricular ejection fraction (LVEF greater than or equal to 55% or normal by NIH Clinical Center criteria).

EXCLUSION CRITERIA:

* Patients who, in the view of the treating physician, have significant active hepatic, renal, pulmonary or psychiatric diseases are ineligible.
* 2 Prior treatment with AZD7451.
* History of hypersensitivity to active metabolites or excipients of AZD7451.
* Clinically significant cardiovascular event (e.g. myocardial infarction, angina pectoris, coronary artery bypass graft, angioplasty, vascular stent, superior vena cava syndrome (SVC), New York Heart Association (NYHA, Appendix I) classification of heart disease >2 within 6 months before entry; or presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
* Hemorrhagic or ischemic stroke, including transient ischemic attacks and other central nervous system bleeding in the preceding 6 months that were not related to glioma surgery. History of prior intratumoral bleeding is not an exclusion criterion; patients with history of prior intratumoral bleeding, however, need to undergo a non-contrast head CT to exclude acute blood.
* Ventricular arrhythmias requiring continuous therapy or asymptomatic sustained ventricular tachycardia within 12 months before study entry. Continuous or intermittent atrial fibrillation requiring treatment. Patients with significant ECG abnormalities such as complete left bundle block and third degree heart block are not eligible.
* QTc prolongation with other medications that required discontinuation of that medication.
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
* QTc with Bazett s correction that is unmeasurable, or >470 msec on screening ECG. (Note: If a subject has a QTc interval >470 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be less than or equal to 470 msec in order for the subject to be eligible for the study. Patients who are receiving a drug that has a risk of QTc prolongation excluded if QTc is greater than or equal to 460 msec.
* Any concurrent medication that may cause QTc prolongation or induce

Torsades de Pointes 1) Drugs listed in Appendix H, Table 2, that in the investigator s opinion cannot be discontinued are allowed; however, must be monitored closely.

* Concomitant medications that are moderate or potent inducers or inhibitors of CYP3A4 are not permitted within the specified wash-out periods prior to or during treatment with AZD7451
* Patients with a history of corneal disease such as corneal ulcers, corneal dystrophies, keratoconus.
* Refractory nausea and vomiting or significant gastrointestinal impairment, as judged by the investigator, that would significantly affect the absorption of AZD7451, including the ability to swallow the oral solution.
* Patients known to have active hepatitis B or C (testing not required for entry on study).
* Other concomitant anti-cancer therapy except corticosteroids.
* Patients with a peripheral neuropathy CTCAE > 1 in the prior 4 weeks or active muscle diseases (including dermatomyositis, polymyositis, inclusion body myositis, muscular dystrophy and metabolic myopathy) or family history of myopathy. Patients with pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi syndrome or renal tubular acidosis.
* Evidence of active infection or active bleeding diatheses.
* Pregnant women are excluded from this study because AZD7451 is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD7451, breastfeeding should be discontinued if the mother is treated with AZD7451. Female patients must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:
* Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
* Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Patients known to have a malignancy (other than their malignant glioblastoma) that has required treatment in the last 12 months and/or is expected to require treatment in the next 12 months (except for non-melanoma skin cancer, carcinoma in situ in the cervix or ductal carcinoma in situ).
* Major surgery within 4 weeks or incompletely healed surgical incision before starting therapy.
* Patients known to be HIV-positive (testing is not required for entry on study) and on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD7451. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10-05; Primary Completion 2014-04-23 (Actual); Study Completion 2014-04-23 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose of AZD7451 on a continuous once daily schedule in patients with recurrent gliomas not on enzyme-inducing anti-epileptic drugs (EIAED). | 3 years

SECONDARY OUTCOMES:
To obain exploratory information about the anti-tumor activity of AZD7451. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Teri N Kreisl, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Scanlon PW, Taylor WF. Radiotherapy of intracranial astrocytomas: analysis of 417 cases treated from 1960 through 1969. Neurosurgery. 1979 Sep;5(3):301-8. PMID 228216
- [Background] FRANKEL SA, GERMAN WJ. Glioblastoma multiforme; review of 219 cases with regard to natural history, pathology, diagnostic methods, and treatment. J Neurosurg. 1958 Sep;15(5):489-503. doi: 10.3171/jns.1958.15.5.0489. No abstract available. PMID 13576192
- [Background] Bloom HJ. Combined modality therapy for intracranial tumors. Cancer. 1975 Jan;35(1):111-20. doi: 10.1002/1097-0142(197501)35:13.0.co;2-#. PMID 162849